CLINICAL TRIAL: NCT02510118
Title: Synergistic Anti-tumor Effect of ChangTai Keli Based on Chemotherapy for Colon Cancer Patients：a Randomized, Parallel-group, Double-blind, Multicenter Clinical Study
Brief Title: Synergistic Anti-tumor Effect of ChangTai Keli for Colon Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing NingQi Medicine Science and Technology Co., Ltd. (Industry)
Collaborators: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BL2014099-Y0103; Y0103 (Registry Identifier: BL2014099)
Record Dates: First submitted 2015-07-12; First posted 2015-07-28 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Colon Cancer
Keywords: ChangTai Keli; Colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — XELOX

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional chemotherapy + placebo ChangTai Keli (Experimental): Patients in this group will be given conventional chemotherapy medicine: modified FOLFOX6 (mFOLFOX6) chemotherapy or XELOX recommended by treatment guidelines for colon cancer, and the placebo ChangTai Keli corresponding to the traditional Chinese syndrome of dampness stasis type of spleen deficiency.
  Interventions: Drug: mFOLFOX6; Drug: XELOX; Drug: Placebo ChangTai Keli
- conventional chemotherapy + ChangTai Keli (Experimental): Patients in this group will be given conventional chemotherapy medicine: modified FOLFOX6 (mFOLFOX6) chemotherapy or XELOX recommended by treatment guidelines for colon cancer, and the ChangTai Keli corresponding to the traditional Chinese syndrome of dampness stasis type of spleen deficiency, a herbal extract twice daily for 26 weeks for lower dosage.
  Interventions: Drug: mFOLFOX6; Drug: XELOX; Drug: ChangTai Keli

INTERVENTIONS:
Drug: mFOLFOX6 — mFOLFOX6 regimen is a combination therapy of oxaliplatin (85 mg/m^2) administered as a 2-hour infusion on Day 1; leucovorin (400 mg/m^2) administered as a 2-hour infusion on Day 1; followed by a loading dose of 5-fluorouracil (5-FU; 400 mg/m^2) IV bolus administered over approximately 2 to 4 minutes on Day 1, then 5- FU (2400 mg/m^2) via ambulatory pump administered for a period of 46 to 48 hours.
Drug: XELOX — XELOX is a combination therapy of Oxaliplatin 130mg/ m^2 d1 Intravenous infusion, every 3 weeks. and Capecitabine 1000mg/m^2 bid, days 1-14, every 3 weeks
Drug: Placebo ChangTai Keli — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of dampness stasis type of spleen deficiency will be given placebo ChangTai Keli, twice daily for 26 weeks for lower dosage.
  Arms: conventional chemotherapy + placebo ChangTai Keli
Drug: ChangTai Keli — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of dampness stasis type of spleen deficiency will be given placebo ChangTai Keli, twice daily for 26 weeks for lower dosage.
  Arms: conventional chemotherapy + ChangTai Keli

SUMMARY:
The aim of this study is to evaluate the synergistic anti-tumor effect of ChangTai Keli based on chemotherapy for colon cancer patients by a randomized, parallel-group, double-blind, multicenter clinical study.

DETAILED DESCRIPTION:
Although many therapies exist and are being developed to relieve symptoms for colon cancer, there are few randomized controlled clinical trials to evaluate comprehensive Traditional Chinese medicine (TCM) interventions in colon cancer. The aim of this study is to evaluate the synergistic anti-tumor effect of ChangTai Keli based on chemotherapy for colon cancer patients. This is a multi-center, randomized, double-blind, placebo-controlled study to evaluate the synergistic anti-tumor effect of TCM on colon cancer patients. Following a run-in period, approximately 360 subjects will be randomly assigned to conventional chemotherapy treatment group, ChangTai Keli and conventional chemotherapy treatment group for 26 weeks. After the 26 weeks treatment period, subjects in two treatments arms will follow-up 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. collaboration from hospital oncology patients in hospital. Confirmed by pathology or cytology for colon cancer, Ⅱ A - Ⅳ period of patients with colon cancer line (or late postoperative palliative chemotherapy).
2. age > 18 years of age, and the 75 - year - old patient or less;
3. fitness score (ECOG PS) 2 minutes or less, expected lifetime > 6 months;
4. volunteered for the clinical research, and sign the informed consent.

Exclusion Criteria:

1. patients with other primary malignant tumors within 1 year;
2. intentional, severe liver and kidney disease patients with serious obstacle and function;
3. pregnancy or lactation women, mental disorders to cooperate to complete the healer;
4. is in other subjects or attended other drugs test interval < 3 months.
5. do not meet the inclusion criteria;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Event (AE) | The time frame for adverse event reporting is from the first dose date to 30 days since the last dose date
  Severity was graded using Common Terminology Criteria for Adverse Events (CTCAE) v3.0, with the exception of some dermatology/skin adverse events that were graded using CTCAE v3.0 with modifications. Fatal adverse events are classified as grade 5. Serious adverse events include any event that is fatal, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or other significant medical hazard. Treatment-related AEs were those that the investigator considered a reasonable possibility that might have been caused by study drug.
Quality of life | Change from Baseline in the QLQ-C30 (V3.0)at the week 2, 4, 6, 8, 10,13, 26 of the treatment phase, the week 13, 26, 39 and 52, 65, 78, 91, 104, 117, 130 of the followup phase.
  Using QLQ-C30 (V3.0) to asses the impact of COPD on a person's life, and how this changes over time.

SECONDARY OUTCOMES:
symptom | Change from Baseline in symptom score at the week 2, 4, 6, 8, 10,13, 26 of the treatment phase, the week 13, 26, 39 and 52, 65, 78, 91, 104, 117, 130 of the followup phase.
  Using TCM scale to assess a patient's level of syptom. The symptom scale is a simple grading system that scored from 0, 2, 4, 6.
Investigator-assessed Progression-Free Survival (PFS) | 3 years
  The time from the date of randomization until objective tumor progression or death due to any cause. Objective tumor progression was determined through radiological imaging and based on the requirements of the Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1)
Progression-free Survival (PFS) | the time from the date of randomization to the date of first disease progression, or death within 60 days after the last evaluable tumor assessment or randomization date (whichever was later)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoning Wang, Professor, Principal Investigator — China:Jiangsu province hospital of integrated traditional Chinese and western medicine
Locations (1):
- Jiege Huo, Nanjing, Jiangsu, China